CLINICAL TRIAL: NCT00000710
Title: A Phase I Safety, Efficacy, and Pharmacokinetic Study of 2',3'-Dideoxyinosine (ddI) Administered Twice Daily to Patients With AIDS or AIDS Related Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 064; 11038 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Injections, Intravenous; Didanosine; Dose-Response Relationship, Drug; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
To determine the safety, pharmacokinetics (blood levels), and effectiveness of didanosine (ddI) when administered both intravenously and orally. After the maximum tolerated dose (MTD) is determined, an appropriate dosage regimen will then be established for Phase II and Phase III trials.

Zidovudine (AZT) has produced the best clinical results in the drug therapy of AIDS to date, but it produces toxicity in approximately 50 percent of patients. Early data show that ddI possesses high antiviral activity and less toxicity than AZT. The most effective route and dose of ddI has yet to be determined.

DETAILED DESCRIPTION:
Zidovudine (AZT) has produced the best clinical results in the drug therapy of AIDS to date, but it produces toxicity in approximately 50 percent of patients. Early data show that ddI possesses high antiviral activity and less toxicity than AZT. The most effective route and dose of ddI has yet to be determined.

Patients are given intravenous drug for 14 days with a 1 day washout period, then 76 weeks of oral medication. To expedite this safety study and still be able to maintain close monitoring of the patient's health, an overlapping dosing regimen is used. After 6 patients have been enrolled and at least 4 have completed 4 weeks of dosing without significant toxic effects, a second group of patients is started at the next dose level.

AMENDED: An alternative oral dosing formulation of ddI will be provided as a buffer powder blend packaged in sealed foil sachets in several strengths.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* Allopurinol for consistent occurrence of hyperuricemia observed with 2',3'-dideoxyinosine (ddI) administration.

Allowed:

* Aerosolized pentamidine for Pneumocystis carinii pneumonia (PCP) prophylaxis.
* Oral acyclovir for herpes simplex infections provided ddI dosing is suspended during this time.
* Ketoconazole for patients not responding to any other therapy and after consultation with the sponsor.
* Symptomatic therapy such as analgesics, antihistamines, antiemetics, antidiarrheal agents, or other supportive therapy may be administered as deemed necessary by the principal investigator.
* Aspirin rather than acetaminophen for fever.

Patients with the following will be included:

* An absence of life-threatening opportunistic infection on enrollment.
* A life expectancy less than 6 months.
* Available for follow-up for at least 6 months.
* Able to provide informed consent. Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Intractable diarrhea.
* No venous access.
* A history of or propensity for seizure disorders.
* A history of past or current heart disease or other significant abnormality on routine EKG.

Concurrent Medication:

Excluded:

* Adenine deaminase inhibitors.
* Trimethoprim / sulfamethoxazole for Pneumocystis carinii pneumonia (PCP) infections.
* Antibiotics.
* Acetaminophen for therapy of fever.

Patients with the following are excluded:

* Intractable diarrhea.
* A life expectancy less than 6 months.
* No venous access.
* A history of or propensity for seizure disorders.
* A history of past or current heart disease or other significant abnormality on routine EKG.

Prior Medication:

Excluded:

* Any agent known as a potent inducer or inhibitor of drug-metabolizing enzymes.
* Excluded within 2 weeks of study entry:
* Trimethoprim / sulfamethoxazole.
* Excluded within 1 month of study entry:
* Any antiretroviral drug.
* Investigational agents.
* 2',3'-didanosine.
* AL721.
* Interferons.
* Immunomodulating drugs.
* Excluded within 3 months of study entry:
* Ribavirin.
* Cytotoxic agents.

Risk Behavior:

Excluded:

Active alcohol or drug abuse sufficient in the investigator's opinion to prevent adequate compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Study Completion 1990-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolin R, Study Chair
Locations (1):
- SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York, United States

REFERENCES:
- [Background] Demeter L, Nawaz T, Morse G, Dolin R, Reichman R. AZT resistant (AZT-R) HIV-1 isolates obtained during DDI monotherapy from a patient with no history of AZT use. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:139
- [Background] Valentine FT, Seidlin M, Hochster H, Laverty M. Phase I study of 2',3'-dideoxyinosine: experience with 19 patients at New York University Medical Center. Rev Infect Dis. 1990 Jul-Aug;12 Suppl 5:S534-9. doi: 10.1093/clinids/12.supplement_5.s534. PMID 1974725
- [Background] Lambert J, Dolin R, Seidlin M, Knupp C, McLaren C, Reichman RC. Phase I study of 2'3'dideoxyinosine(ddI) administered twice daily to patients with AIDS/AIDS related complex. Int Conf AIDS. 1989 Jun 4-9;5:563 (abstract no MCP130)
- [Background] Seidlin M, Lambert JS, Dolin R, Valentine FT. Pancreatitis and pancreatic dysfunction in patients taking dideoxyinosine. AIDS. 1992 Aug;6(8):831-5. doi: 10.1097/00002030-199208000-00011. PMID 1418780
- [Background] Lambert JS, Seidlin M, Valentine FT, Reichman RC, Dolin R. Didanosine: long-term follow-up of patients in a phase 1 study. Clin Infect Dis. 1993 Feb;16 Suppl 1:S40-5. doi: 10.1093/clinids/16.supplement_1.s40. PMID 8093846
- [Background] Dolin R, Lambert JS, Morse GD, Reichman RC, Plank CS, Reid J, Knupp C, McLaren C, Pettinelli C. 2',3'-Dideoxyinosine in patients with AIDS or AIDS-related complex. Rev Infect Dis. 1990 Jul-Aug;12 Suppl 5:S540-9; discussion S549-51. PMID 1974726
- [Background] Lambert JS, Seidlin M, Reichman RC, Plank CS, Laverty M, Morse GD, Knupp C, McLaren C, Pettinelli C, Valentine FT, et al. 2',3'-dideoxyinosine (ddI) in patients with the acquired immunodeficiency syndrome or AIDS-related complex. A phase I trial. N Engl J Med. 1990 May 10;322(19):1333-40. doi: 10.1056/NEJM199005103221901. PMID 2139173
- [Background] Demeter LM, Nawaz T, Morse G, Dolin R, Dexter A, Gerondelis P, Reichman RC. Development of zidovudine resistance mutations in patients receiving prolonged didanosine monotherapy. J Infect Dis. 1995 Dec;172(6):1480-5. doi: 10.1093/infdis/172.6.1480. PMID 7594706
- [Background] Kieburtz KD, Seidlin M, Lambert JS, Dolin R, Reichman R, Valentine F. Extended follow-up of peripheral neuropathy in patients with AIDS and AIDS-related complex treated with dideoxyinosine. J Acquir Immune Defic Syndr (1988). 1992;5(1):60-4. PMID 1346633